CLINICAL TRIAL: NCT05748782
Title: Efficiency and Safety of BASKA Mask Ventilation in Comparison With Endotracheal Intubation During Otologic Surgery in the Lateral Head and Neck Position
Brief Title: BASKA Mask in Otologic Surgery in Lateral Position
Acronym: BASKAvsETT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, professor, Assiut University
Other Study IDs: BASKA mask in otologic surgery
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Airway Device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BASKA GROUP: the BASKA mask will be inserted, and its size will be chosen according to the manufacturer's weight-based recommendations.
  Interventions: Other: Baska Mask
- ETT GROUP: Patients in this group will be anesthetized using an endotracheal tube of appropriate size.
  Interventions: Device: Endotracheal tube

INTERVENTIONS:
Other: Baska Mask — The Baska mask (Logikal Health Products PTY Ltd., Morisset, NSW, Australia) is a supraglottic airway device introduced in 2012 with many innovations that might be expected to overcome these derangements.
  Groups: BASKA GROUP
Device: Endotracheal tube — BASKA Mask
  Other Names: ETT
  Groups: ETT GROUP

SUMMARY:
This study aims to evaluate the Efficiency and safety of BASKA mask ventilation in comparison with endotracheal intubation during otologic surgery performed with the head and neck in the lateral position. The primary outcome will be the intraoperative peak inspiratory pressure (PIP). Secondary outcomes will be intraoperative lung mechanics, oropharyngeal leak pressure (OLP), ventilation score, fiberoptic glottic view score, and perioperative adverse effects.

DETAILED DESCRIPTION:
The laryngeal mask airway (LMA) was invented in 1981 by Dr Brain Because of its advantages, LMAs are increasingly used as a substitute for endotracheal tubes in a variety of surgical situations requiring general anesthesia. With the appearance of various new LMAs that address the limitations of the classic model, not only has their use in selective operations increased, but the indications for LMA have also grown LMAs can be inserted into the hypopharynx easily without laryngoscopy and neuromuscular blocking agents, and they can also be removed from the patient's mouth quickly. Decreasing airway irritation during surgery results in fewer hemodynamic changes and airway accidents from anesthesia and enables wakeup with less coughing and bucking, which could result in less ossicular replacement prosthesis displacement .

In middle ear/mastoid procedures, because the operation involves the temporal bone, including the surrounding normal nerves and blood vessels, improper manipulation can lead to complications such as facial paralysis; therefore, the operation needs to be performed carefully. Compared to endotracheal intubation, LMAs have little effect on middle ear pressure . These advantages make anesthesiologists prefer LMAs during otologic surgery. In addition, since LMAs can reduce the response to upper airway stimulation, they can be used as an airway device during surgery requiring facial nerve monitoring without the use of muscle relaxants .

However, the points of contention and primary disadvantages of the use of LMA are the reduced levels of airway protection, the increased risk of gastric insufflation, the difficulty of insertion, partial upper airway obstruction and the possibility of dislocation during the procedure . To expose the operative field, otologists usually require the patient's head be rotated 60°~90° to the healthy side. Some studies have reported that the head and neck position can affect the sealing and ventilation functions of LMAs and the fiberoptic view .

The Baska mask (Logikal Health Products PTY Ltd., Morisset, NSW, Australia) is a supraglottic airway device introduced in 2012 with many innovations that might be expected to overcome these derangements . First, its' non-inflatable cuff is continuous with the central channel of the device and automatically inflates during positive pressure ventilation in response to the increased inflation pressure. This inflation produces an oropharyngeal leak pressure higher than that produced by other LMAs, enabling more effective ventilation. Second, it has an esophageal drainage inlet and side channels that comprise an efficient pharyngeal drainage system which facilitates aspiration of gastric contents, thereby reducing the risk of gastric overinflation and pulmonary aspiration. Third, a strong integrated bite-block that acts as a safeguard against obstruction of the Baska mask.

In this study, the hypothesis is that these modifications might enable the Baska mask to become a reasonable and safe alternative to the endotracheal intubation in during otologic surgery performed with the head and neck in the lateral position.

ELIGIBILITY:
Inclusion Criteria:

1. Age group 18 - 60 years old.
2. Both genders.
3. Undergoing general anesthesia for ear surgeries in the lateral neck position (60-90 degrees) in whom BASKA mask can be a suitable device for airway management

Exclusion Criteria:

1. Patient refusal,
2. History of cardiac or respiratory disease, psychological disorders,
3. High risk of regurgitation or aspiration based on a history of diabetes, hiatus hernia, gastroesophageal reflux, and obesity,
4. neck pathology,
5. Predicted difficult airway (history of difficult airway, mouth opening <2.5cm, Modified Mallampati class III/IV, thyro-mental distance <6.5cm or cervical spine pathology),

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients Undergoing general anesthesia for ear surgeries in the lateral neck position (60-90 degrees) in whom BASKA mask can be a suitable device for airway management.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-23 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the intraoperative peak inspiratory pressure (PIP) | Intraoperative
  the peak inspiratory pressure will be measured from the panel of the ventilator electronic box (Datex-Ohmeda,Inc 3030 Ohmeda Drive PO Box 7550 )

SECONDARY OUTCOMES:
Oropharyngeal leak pressure | Intraoperative
  The fresh gas flow will be adjusted to 3 l/min, and the electronic APL valve is set automatically at 30 cmH2O, the airway pressure rises until attaining a plateau that is equal to the total leak pressure of the LMA with an upper limit of airway pressures 40 cm H2O. The airway pressure at which an audible leak is detected at the mouth and auscultated by placing the stethoscope over the patient's neck just lateral to the thyroid cartilage will be recorded as the oropharyngeal leak pressure (OLP) .
Ventilation Score | Intraoperative
  The ventilation score which will be scored from 0 to 3 based on three criteria: no leakage with an airway pressure of 15 cm H2O, bilateral chest excursions with a peak inspiratory pressure of 20 cm of H2O, and a square wave capnography, with each item scoring 0 or 1 point.
Fiberoptic Glottic Score | Intraoperative
  position of the device concerning the glottis will be investigated by inserting a fiberoptic laryngoscope (11301BNX, diameter 5.5 mm; length 65 cm; Karl Storz, Tuttlingen, Germany) will be inserted through the mask to evaluate the glottic view. Oxygen will be administered through the suction port throughout the procedure. Fiberoptic images will be graded with Brimacombe score that ranges from one to five; (grade1= only larynx seen, grade 2=larynx and epiglottis posterior surface seen, grade 3=larynx and epiglottis tip of anterior surface seen, 50% visual obstruction of epiglottis to larynx and grade 5, i.e. epiglottis down folded and larynx cannot be seen directly.

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — Assiut University
Locations (1):
- Main Assiut University Hospital, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No